CLINICAL TRIAL: NCT01337245
Title: Emergency Treatment of Coral Snake Envenomation With Antivenom
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS-02/08; FD003706 (Other Grant/Funding Number: FDA OOPD)
Record Dates: First submitted 2011-04-15; First posted 2011-04-18 (Estimated); Results first posted 2023-04-05 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Coral Snake Bite; Toxic Effect of Coral Snake Venom
Keywords: Envenomation; Coral Snake; Antivenom; Micrurus fulvius

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Antivenom (Experimental): For comparison with historical mortality rate, all patients prospectively enrolled will receive antivenom (Snake [Micrurus] North American immune F(ab')2 Equine) for treatment of coral snake bite.
  Interventions: Drug: Snake (Micrurus) North American immune F(ab')2 Equine

INTERVENTIONS:
Drug: Snake (Micrurus) North American immune F(ab')2 Equine — 5 vials of study drug reconstituted and diluted to 250 mL Normal Saline and administered intravenously.

SUMMARY:
The purpose of this study is to see whether a new F(ab')2 antivenom will prevent injury and death from the bite of a coral snake.

Funding Source - FDA OOPD.

DETAILED DESCRIPTION:
Coral snake bites may be trivial in effect, or they may cause profound and life-threatening respiratory paralysis, depending on the severity of the envenomation. Venom toxins target the neuromuscular junction, where effects typically become apparent hours following the bite, by which time the clinical syndrome may be irreversible. Unless neurotoxicity is prevented, ventilatory paralysis may cause death or require intensive care for weeks after the bite. Prevention of paralysis, historically, has involved treating all bite victims with antivenom.

This protocol will enable the therapeutic use of a new F(ab')2 antivenom in the management of coral snake envenomation.

Following a coral snake bite, patients who meet inclusion/exclusion criteria and who provide informed consent will receive 5 vials of antivenom intravenously over no less than 30 minutes. Blood assays for venom levels and clinical assessments of neurologic status before and after treatment will be conducted and patients will be followed for 22 days for safety and survival endpoints.

The primary endpoint of this Phase 3 trial will be survival, for comparison with a historical mortality rate of 15%.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of any age. Presenting for emergency treatment of coral snake bite.

Exclusion Criteria:

* Prior use of coral snake antivenom for this envenomation. Allergy to horse serum.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-05; Primary Completion 2016-11-11 (Actual); Study Completion 2016-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Boyer, MD, Study Director — VIPER Institute, University of Arizona; Jason W. Wilson, MD, Principal Investigator — Tampa General Hospital
Locations (5):
- United States (5):
  - Banner University Medical Center, Tucson, Arizona
  - Florida Hospital Deland, DeLand, Florida
  - Lee Memorial Hospital, Fort Myers, Florida
  - St. Lucie Medical Center, Port Saint Lucie, Florida
  - Tampa General Hospital, Tampa, Florida

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Antivenom
Started | 26
Completed | 25
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Antivenom
Number analyzed (Participants) | 26
Age, Continuous [Mean (Full Range); unit: years] | 39.7 [11 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 23
  Race/Ethnicity: Black | 1
  Race/Ethnicity: Hispanic | 1
  Race/Ethnicity: Unknown | 1
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Survived
Time Frame: Immediately following start of infusion (day 1) through Day 22
Measure: Count of Participants; unit: Participants
Arm/Group | Antivenom
Number analyzed (Participants) | 25
Participants | 25

2. Secondary Outcome: Change in Mean Venom Level From Baseline to 24 Hours
Time Frame: Through 24 hours
Population: Subjects with blood successfully collected at 24 hours
Measure: Mean (Full Range); unit: ng per ml
Arm/Group | Antivenom
Number analyzed (Participants) | 23
ng per ml | -34.5 [-353 to 0]

3. Secondary Outcome: Change in Mean Antivenom Level From Baseline to 24 Hours
Time Frame: Through 24 hours
Measure: Mean (Full Range); unit: mcg per ml
Arm/Group | Antivenom
Number analyzed (Participants) | 23
mcg per ml | 112.4 [62.6 to 236.4]

ADVERSE EVENTS:
Time Frame: 22 Days
Arm/Group | Antivenom
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 3/26
Other Adverse Events (participants affected / at risk) | 23/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antivenom (N=26)
Type I immediate hypersensitivity reaction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hospital Re-admission (Infections and infestations) | 1 (1) — Cellulitis
Alcohol withdrawal resulting in prolonged hospitalization (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antivenom (N=26)
Rash (Skin and subcutaneous tissue disorders) | 6 (6)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Forgetfulness (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Runny nose (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Lightheadedness (Nervous system disorders) | 2 (2)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 5 (8)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Acute immune reaction (Immune system disorders) | 6 (8)
Laceration (Skin and subcutaneous tissue disorders) | 1 (1)
Spider bite (Skin and subcutaneous tissue disorders) | 1 (1)
Numbness (Skin and subcutaneous tissue disorders) | 2 (2)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Local swelling (Skin and subcutaneous tissue disorders) | 4 (4)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 1 (1)
Hyperesthesia (Skin and subcutaneous tissue disorders) | 1 (1)
Blurry vision (Eye disorders) | 1 (1)
Redness of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 2 (2)
Swollen lymph node (Immune system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Swollen lips (Skin and subcutaneous tissue disorders) | 1 (1)
Ethanol withdrawal (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes